CLINICAL TRIAL: NCT03959722
Title: The Effect of Probiotics on the Relationship Between the Gut Microbiota and Gastrointestinal Symptoms During Endurance Exercise'
Brief Title: The Effect of Probiotics on GI Symptoms
Acronym: WHOMLF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Karlijn te Poele (Other)
Collaborators: VU University of Amsterdam (Other); Wageningen University and Research (Other); Universiteit Leiden (Other); MyMicroZoo (Unknown); Winclove Bio Industries BV (Industry)
Responsible Party: Sponsor-Investigator, Karlijn te Poele, MSc., Hogeschool Leiden, University of Applied Science
Organization: Hogeschool Leiden, University of Applied Science (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NL69974.081.19
Record Dates: First submitted 2019-05-14; First posted 2019-05-22 (Actual); Last update posted 2020-09-09 (Actual); Status verified 2020-09

CONDITIONS: Gastrointestinal Symptoms
Keywords: Endurance athletes; probiotics; endurance exercise

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Probiotics:Healthy male endurance athletes with GI symptoms (Experimental): 14 weeks of supplementation with a multispecies probiotics: Ecologic® PERFORMANCE ( 1*1010 CFU(Colony forming units)/daily dose, Winclove Probiotics B.V., Amsterdam).
  Interventions: Dietary Supplement: Ecologic® PERFORMANCE
- Placebo: Healthy male endurance athletes with GI symptoms (Placebo Comparator): 14 weeks of supplementation with a placebo comparator (Winclove Probiotics B.V., Amsterdam)
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Ecologic® PERFORMANCE — Ecologic® PERFORMANCE is a probiotic formulation consisting of different probiotic bacterial strains, namely:
  Bifidobacterium bifidum W23 Bifidobacterium lactis W51 Enterococcus faecium W54 Lactobacillus acidophilus W22 Lactobacillus brevis W63 Lactococcus lactis W58
  Except for the bacterial strains, Ecologic® PERFORMANCE contains the following other ingredients:
  * maize starch and maltodextrins
  * fructo-oligosaccharides (FOS) P6 and Polydextrose P4 (strain specific prebiotics)
  * vegetable protein
  * mineral mix (Potassium chloride, Magnesium sulphate, Manganese sulphate)
  Arms: Probiotics:Healthy male endurance athletes with GI symptoms
Dietary Supplement: Placebo — The placebo contains no bacterial strains, but the following ingredients:
  * maize starch and maltodextrins
  * fructo-oligosaccharides (FOS) P6 and Polydextrose P4 (strain specific prebiotics)
  * vegetable protein
  * mineral mix (Potassium chloride, Magnesium sulphate, Manganese sulphate)
  Arms: Placebo: Healthy male endurance athletes with GI symptoms

SUMMARY:
A double-blind randomized, placebo-controlled study will be performed with experienced endurance athletes to assess the effect of probiotics supplementation on the occurrence and intensity of the gastrointestinal symptoms, on performance and on the composition and function of the gut microbiota. The duration of the supplementation period, with Ecologic® PERFORMANCE supplements, is fourteen weeks. Standardized maximum exercise tests on a treadmill are performed before and after the supplementation period, as well as two performance tests (before) and one performance test (after). During the performance tests, the load is first submaximal for 1 hour, after which a time trial of 30 minutes will be performed. The measurements before and after the supplementation period are performed on individual days with at least 48 hours of relative rest in between. During the supplementation period, training diaries, a Profile of Mood States (POMS) questionnaire and a few questionnaires about dietary habits will be completed.

DETAILED DESCRIPTION:
Rationale: Endurance exercise, such as running a marathon, is becoming increasingly popular. In addition to the many positive health effects of endurance exercise, it can also be accompanied by gastrointestinal symptoms. For example, around 30-90% of runners suffer from gastrointestinal symptoms during or in the hours after intensive/endurance running. The occurrence of gastrointestinal symptoms is probably due to the redistribution of blood volume, resulting in less blood supply to the digestive tract and a less functioning intestinal barrier. Because the intestinal barrier functions less, endotoxins can enter the bloodstream and cause inflammatory reactions. Running in the heat causes extra redistribution of the blood volume, because extra blood is needed for cooling of the body. It is known that the gut microbiota affect food digestion, but also the functioning of the cells that line the intestinal wall and the connections between these cells. It is possible that runners with gastrointestinal symptoms face a different composition of the gut microbiota and / or metabolites during endurance exercise compared to runners without any complaints, as a result of which the gut barrier functions less well and problems may occur. Many positive effects have been attributed to the use of probiotics in general. Amongst which, the reduction of gastrointestinal symptoms during endurance exercise, probably due to improvement in intestinal permeability. Hence, the main goal of our research project is to investigate whether the chance of and/or intensity of gastrointestinal symptoms during endurance exercise and the exercise performance can be influenced by probiotics supplementation in trained endurance athletes. This will be studied in relation to the composition of the gut microbiota and / or metabolites.

Objective:

Primary Objective:

Can the chance at and/or intensity of gastrointestinal symptoms during exercise be influenced by probiotics supplementation in trained endurance athletes who experience these symptoms and can performance be enhanced? Secondairy Objective: Can the composition and function of the gut microbiota of trained athletes that experience gastrointestinal symptoms during exercise be positively influenced by probiotics supplementation?

Study design: A double-blind randomized placebo-controlled trial will be performed to investigate the effect of 14 weeks probiotics supplementation with Ecologic® PERFORMANCE supplements. Standardized maximal incremental exercise tests will be performed before and after the supplementation period, as well as two performance tests (before) and one performance test (after). During the supplementation period training diaries, a POMS questionnaire and some questionnaires about food habits will be completed, a food diary and Food Frequency Questionnaire (FFQ).

Study population: Healthy male endurance athletes of Dutch nationality, 18-45 years old, who regularly experience gastrointestinal symptoms during exercise.

Intervention: Fourteen weeks of supplementation with Ecologic® PERFORMANCE probiotics supplements (or placebo).

Main study parameters/endpoints: Main study endpoints are differences in changes in the severity and occurrence of gastrointestinal symptoms and changes in exercise performance (total distance on a time trial and maximum speed during an incremental exercise test). Also changes in composition of the microbiota and differences in changes in the metabolites in the stool sample before and after the supplementation period in the experimental and control group will be studied.

Nature and extent of the burden and risks associated with participation, benefit and group relatedness: Benefits will be the value of the test results and outcome measures of the microbiome analysis. Also the chance on a reduced risk of occurrence of gastrointestinal symptoms might be of value for potential participants. The risks for the participants are minor. Only participants that are healthy and endurance trained will be included. In the Human Performance Laboratory of the Faculty of Behavioural and Human Movement Sciences, performance tests in warm conditions are executed regularly and health risks related to the experimental protocol are minor for the participants since they are already well-trained and the exercise intensity will be relatively well-tolerated, since they are used to similar efforts. Probiotics supplements are freely available at the market, and the Ecologic® PERFORMANCE supplements are available in the web shop of Winclove B.V. The same supplement has been used before in the same dosage and no adverse effects were reported. Participants will fill in a food frequency questionnaire and questionnaire about gastrointestinal symptoms and hand in a stool sample before and after the supplementation period. They will be asked to maintain a training diary during the supplementation period and also fill in the POMS questionnaire weekly. The maximal incremental exercise test (2 times) consists of a warming-up followed by incremental increase in running velocity until voluntary exhaustion. The performance tests (3 times) consists of 60 minutes of submaximal running followed by a time trial of 30 minutes in which participants need to accomplish as much distance as possible.

ELIGIBILITY:
Inclusion Criteria:

* Dutch nationality; maximal oxygen uptake (V ̇O_2max) ≥ 45 mL·kg-1·min-1 (based on an incremental exercise test you are considered trained);
* an average training frequency of at least three times per week;
* a low risk profile based on a health-history form (the form is attached to the participant information letter);
* occurrence of exercise-induced gastrointestinal symptoms.

Exclusion Criteria:

* smoking;
* a diagnosis of gastrointestinal disorders (e.g. Crohn's disease, celiac disease, diagnosed with irritable bowel syndrome);
* use of antidepressants in the 6 months prior to the start of the study;
* use of antibiotics, antivirals, antifungals, antiparasitic agents, prebiotics/probiotics supplements (foods are allowed) in the 6 months prior to the start of the study.

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 42 (Actual)
Dates: Start 2019-11-19 (Actual); Primary Completion 2020-05-02 (Actual); Study Completion 2020-05-02 (Actual)

PRIMARY OUTCOMES:
Performance maximal running | Before and after 14 weeks of supplementation
  Distance in km on a 30 minute running time trial, preceded by two times 30 minutes submaximal exercise.
Performance maximal running maximal incremental exercise test | Before and after 14 weeks of supplementation
  Maximum speed on a maximal rincremental exercise test
Gastrointestinal symptoms | Before and after 14 weeks of supplementation
  Severity (scale 1-10) of gastrointestinal symptoms during and directly after a running performance test. (1 = none and 10 = worst symptoms ever)

SECONDARY OUTCOMES:
The influence of probiotics on the composition of the gut microbiota in trained endurance athletes that experience gastrointestinal symptoms. | Before and after 14 weeks of supplementation
  Differences in changes in composition of the gut microbiota in the stool sample.
The influence of probiotics on the composition of the gut metabolites in trained endurance athletes that experience gastrointestinal symptoms. | Before and after 14 weeks of supplementation
  Differences in changes in the gut metabolites in the stool sample

OTHER OUTCOMES:
Temperature | Before and after 14 weeks of supplementation
  Body temperature in degrees celcius during endurance exercise, calculated by core temperature and skin temperature
Training diary | During the 14 weeks supplementation period
  Training load (in arbitrary units) calculated by modality, training volume (in km), training intensity (average HR) and a subjective measure of training intensity perception (RPE-scale 1=very, very light -10=maximum)
Profile of Mood States Questionnaire | During the 14 weeks supplementation period
  Summed outcome score of the weekly completed Profile Of Mood States questionnaire (with 32 questions with scale 0-4; 0=not at all - 4=extremely).

CONTACTS AND LOCATIONS:
Overall Officials: Karlijn te Poele, MSc, Principal Investigator — Hogeschool Leiden, University of Applied Sciences
Locations (1):
- Vrije Universiteit Amsterdam, Amsterdam, Netherlands

IPD SHARING:
Plan to Share IPD: No